CLINICAL TRIAL: NCT00324701
Title: Telepsychology-Service Delivery for Depressed Elderly Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other); University of Maryland (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 04-421; HR16402 (Other: Medical University of South Carolina)
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-09

CONDITIONS: Depression; Elderly
Keywords: Mental Health; Geriatric Medicine; Depression; Health Service Delivery; Aged
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Mental Health Teletherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telepsychology (Experimental): therapy done at patients house
  Interventions: Behavioral: Telepsychology
- Face-to-face therapy (Active Comparator): therapy delivered at the VAMC
  Interventions: Behavioral: Face-to-face therapy

INTERVENTIONS:
Behavioral: Telepsychology — therapy done at patients house
  Arms: Telepsychology
Behavioral: Face-to-face therapy — therapy delivered at the VAMC
  Arms: Face-to-face therapy

SUMMARY:
The purpose of this study is to see whether therapy for elderly adults with major depression can be delivered effectively using videoconferencing technology ("telepsychology"), which allows a therapist and patient who are not in the same room as one another to communicate. We are interested in learning if this form of mental health service delivery is an acceptable alternative to traditional face-to-face therapy delivered with the therapist in the same room as the patient.

DETAILED DESCRIPTION:
ABSTRACT

Telepsychology: Service Delivery for Depressed Elderly Veterans

1. Objective: The immediate objective is to test the hypothesis that a novel mode of geriatric mental health service delivery, using in-home videoconferencing technology ("Telepsychology"), will be as effective as the traditional mode of service delivery ("Same-Room") for treating older adult veterans suffering from major depressive disorder (MDD). The ultimate objective is to help the VA develop and evaluate strategies for providing mental health care to elderly veterans who live in rural areas, many of whom are minorities.
2. Research Design: This project is a 4-year prospective, randomized between-groups study comparing the efficacy of an intervention for geriatric depression delivered via two different modes (Telepsychology, Same-Room). Participants in the Telepsychology condition will receive care in their own home via videophone contact with a therapist at the Charleston VA Medical Center; participants in the Same-room condition will receive their care via traditional face-to-face therapy sessions held at the Charleston VA Medical Center. Two-hundred twenty-four (224) participants will be recruited from primary care and mental health clinics within the Charleston VA Medical Center catchment area. Treatment will be administered over an 8-week period (active treatment phase); and participants will be followed for an additional 12-months (follow-up phase) to ascertain longer-term effects of treatment on three outcome domains: (1) clinical outcomes: symptom severity and social functioning; (2) process outcomes: patient satisfaction and acceptance, treatment credibility, session attendance, treatment adherence, and treatment dropout; and (3) cost-effectiveness.
3. Methodology: Population and Sample: Participants will be elderly veterans (N = 224), age 60 and above, with diagnoses of major depressive disorder (MDD). Based on our previous research and local demographics, we expect approximately 40% of our sample will be African-American. Types of Data: To assess outcome, we will use measures that have been widely validated in the clinical evaluation of older adults with MDD. Measures will be collected at pre-treatment, post-treatment, 3-, and 12-month follow-up. Data Analyses Plan: The primary clinical response variable is proportion (%) of patients who respond to treatment, where treatment response is defined as at least a 50% improvement from baseline to post-treatment level on the GDS (percent change from baseline:[baseline-post]/baseline >= 50%). Two approaches to estimation of the primary response variable will be taken. The first approach will estimate proportion of responders (% responders) at the end of the 8-week active treatment course based on the total number randomized to each treatment. This is equivalent to a "worst case" analysis in which all premature exits (for whom response status is missing) will be treated as non-responders. We will also estimate proportion of responders for each treatment based on only those who complete the 8-week treatment course (completer analysis). The second approach will use multivariable logistic regression to estimate adjusted % responders. Finally, we will conduct a range of analyses between African-American and Caucasian subjects to look at differential efficacy, patient preferences and satisfaction, and adherence across racial groups.
4. Findings: Analysis of data is currently in process.
5. Clinical Relationship: Findings will allow for improved service delivery and access to elderly depressed veterans.
6. Impact/Significance: The telepsychology literature is undeveloped. The VA has made telehealth a priority strategy for bringing quality services to veterans in rural areas. Therefore, research that addresses the efficacy of this mode of service delivery is acutely needed. If Telepsychology efficacy and cost-effectiveness is demonstrated, then future research and program development will bring specialized mental health services to the homes of minority veterans or VA community based outpatient clinics. Further, if Telepsychology effectiveness can be empirically established, then we can proceed with research that examines a range of important system issues. Thus, this project represents a step in a major programmatic line of research in mental health service delivery to rural and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be older male and female veterans,
* age 60 and above,
* with diagnoses of major depressive disorder (MDD) assigned on the basis of the Structured Clinical Interview for DSM-IV (SCID; Spitzer et al., 1997).

Exclusion Criteria:

* Actively psychotic or demented persons,
* individuals with both suicidal ideation and clear intent, and
* individuals meeting criteria for substance dependence will be excluded from participation.

However, in order to maximize generalization of results, presence of other forms of psychopathology will not be a basis for exclusion. All of these structured interviews will be audiotaped in order to calculate inter-rater reliability on a randomly selected 20%. (See Human Subjects for procedures in place for suicidal participants or potential participants).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2006-09; Primary Completion 2011-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E. Egede, MD MS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

REFERENCES:
- [Background] Cluver JS, Schuyler D, Frueh BC, Brescia F, Arana GW. Remote psychotherapy for terminally ill cancer patients. J Telemed Telecare. 2005;11(3):157-9. doi: 10.1258/1357633053688741. PMID 15901444
- [Result] Egede LE, Frueh CB, Richardson LK, Acierno R, Mauldin PD, Knapp RG, Lejuez C. Rationale and design: telepsychology service delivery for depressed elderly veterans. Trials. 2009 Apr 20;10:22. doi: 10.1186/1745-6215-10-22. PMID 19379517
- [Result] Richardson LK, Frueh BC, Grubaugh AL, Egede L, Elhai JD. Current Directions in Videoconferencing Tele-Mental Health Research. Clin Psychol (New York). 2009 Sep 1;16(3):323-338. doi: 10.1111/j.1468-2850.2009.01170.x. PMID 20161010
- [Result] Osborn CY, Egede LE. The relationship between depressive symptoms and medication nonadherence in type 2 diabetes: the role of social support. Gen Hosp Psychiatry. 2012 May-Jun;34(3):249-53. doi: 10.1016/j.genhosppsych.2012.01.015. Epub 2012 Mar 7. PMID 22401705
- [Result] Tuerk PW, Gros DF, Acierno RE, Strachan MK, Egede LE, Morland LA, Greene CJ, Myrick DL, Frueh BC. Delivery of evidence-based psychotherapy via video telehealth. Journal of psychopathology and behavioral assessment. 2013 Dec 1; 35(4):506-521.
- [Derived] Egede LE, Dismuke CE, Walker RJ, Acierno R, Frueh BC. Cost-Effectiveness of Behavioral Activation for Depression in Older Adult Veterans: In-Person Care Versus Telehealth. J Clin Psychiatry. 2018 Aug 28;79(5):17m11888. doi: 10.4088/JCP.17m11888. PMID 30192446
- [Derived] Egede LE, Acierno R, Knapp RG, Walker RJ, Payne EH, Frueh BC. Psychotherapy for Depression in Older Veterans Via Telemedicine: Effect on Quality of Life, Satisfaction, Treatment Credibility, and Service Delivery Perception. J Clin Psychiatry. 2016 Dec;77(12):1704-1711. doi: 10.4088/JCP.16m10951. PMID 27835713
- [Derived] Egede LE, Acierno R, Knapp RG, Lejuez C, Hernandez-Tejada M, Payne EH, Frueh BC. Psychotherapy for depression in older veterans via telemedicine: a randomised, open-label, non-inferiority trial. Lancet Psychiatry. 2015 Aug;2(8):693-701. doi: 10.1016/S2215-0366(15)00122-4. Epub 2015 Jul 16. PMID 26249300

RESULTS

PARTICIPANT FLOW:
Groups:
- Telepsychology: therapy done at patients house using in-home video conferencing technology
- Face-to-face Therapy: therapy delivered at the VAMC in the same room as the therapist
Period: Overall Study
Arm/Group | Telepsychology | Face-to-face Therapy
Started | 120 | 121
Week 8 Assessment | 108 | 107
Completed | 100 | 104
Not Completed | 20 | 17

BASELINE CHARACTERISTICS:
Population: Older adult Veterans (age 60 or older) presenting for services at VA primary care clinics and meeting DSM-IV criteria for major depressive disorder.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telepsychology | Face-to-face Therapy | Total
Number analyzed (Participants) | 120 | 121 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (4.4) | 64.2 (5.6) | 63.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 116 | 119 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 45 | 94
  White | 68 | 75 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Education [Mean (Standard Deviation); unit: years] | 13.5 (2.3) | 13.8 (2.9) | 13.7 (2.6)
Income [Number; unit: participants] — Not all participants answered the question, which explains the discrepancy in total number
  participants
    $0 - < $15,000 | 25 | 24 | 49
    $15,000 - < $25,000 | 24 | 32 | 56
    $25,000 - < $$50,000 | 49 | 44 | 93
    $50,000 or more | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: At Least a 50% Improvement From Baseline to Post-treatment on the Geriatric Depression Scale (GDS)
Description: The Geriatric Depression Scale (GDS) is a 30-item self-report assessment designed specifically to identify depression in the elderly. Participants are asked to respond by answering yes or no in reference to how they felt over the past week. Higher scores indicate more severe depression.
Time Frame: 8 week & 12 months
Population: Participants completing 8 week and 12 month assessments.
Measure: Number (95% Confidence Interval); unit: % participants with treatment response
Arm/Group | Telepsychology | Face-to-face Therapy
Number analyzed (Participants) | 108 | 107
% participants with treatment response
  8 weeks | 17.6 [11.6 to 23.6] | 22.4 [15.8 to 29.1]
  12 months | 22.0 [15.2 to 28.8] | 20.2 [13.7 to 26.7]

2. Secondary Outcome: SCID: Structured Clinical Interview for the DSM-IV
Description: Structured clinical interview for the DSM-IV (SCID) administered by raters blind to subject condition. Structured interviews included psychiatric assessment for depression, PTSD, panic, generalized anxiety disorder (GAD) evaluated using the DSM-IV.
Time Frame: 12 months
Population: Participants completing 12 month assessment
Measure: Number (95% Confidence Interval); unit: % participants with treatment response
Arm/Group | Telepsychology | Face-to-face Therapy
Number analyzed (Participants) | 100 | 104
% participants with treatment response | 50 [41.8 to 58.2] | 44.2 [36.2 to 52.2]

ADVERSE EVENTS:
Arm/Group | Telepsychology | Face-to-face Therapy
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/121
Other Adverse Events (participants affected / at risk) | 0/120 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes